CLINICAL TRIAL: NCT03810573
Title: A Multi-Center, Prospective, Parallel Group, Randomized, Pilot Study Evaluating Safety And Preliminary Effectiveness Of NB1 Bone Graft In Subjects With Degenerative Disc Disease Undergoing Transforaminal Lumbar Interbody Fusion
Brief Title: Evaluation of NB1 Bone Graft Following Lumbar Interbody Arthrodesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bone Biologics Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB1-100
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- NB1-1.5 (Experimental): NB1 low dose
  Interventions: Device: NB1
- NB1-2.0 (Experimental): NB1 high dose
  Interventions: Device: NB1
- Autograft (No Intervention): Autograft

INTERVENTIONS:
Device: NB1 — rhNELL-1/DBX
  Arms: NB1-1.5; NB1-2.0

SUMMARY:
The objective of this clinical study is to evaluate the safety and effectiveness of NB1 Bone Graft in subjects with degenerative disc disease undergoing transforaminal lumbar interbody fusion.

It is estimated that up to 30 participants will be enrolled in approximately 3 clinical sites. During baseline and follow-up assessments, patients will be asked to undergo x-rays and CT scans; adverse events and immunology will be collected, and; participants will be requested to complete participant questionnaires regarding quality of life, pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of degenerative disc disease
* Up to Grade I spondylolisthesis
* Eligible to undergo a single vertebral level spine fusion (L2 to S1)

Exclusion Criteria:

* Previous spinal instrumentation or previous interbody fusion procedure at the involved level
* Grade II or greater spondylolisthesis
* Systemic or local infection at the site of surgery

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Fusion | 12 months
  Defined by an independent (blinded to treatment) radiological assessment as less than five degrees angular vertebral motion, less than three millimeters of translational movement and evidence of bridging bone between the involved vertebral endplates based on x-rays at 12 months after surgery

SECONDARY OUTCOMES:
Removal, revision, or supplemental fixation | 12 months
  Whether there was removal, revision or supplemental fixation of the graft material that required reoperation at the index level during the follow-up period of the study

CONTACTS AND LOCATIONS:
Overall Officials: Tony Goldschlager, MD, Principal Investigator — Monash Health
Locations (3):
- Australia (3):
  - Monash Medical Center, Clayton, Victoria
  - St Vincent Melbourne, Fitzroy
  - St George Hospital, Kogarah

IPD SHARING:
Plan to Share IPD: Yes
As requested
Supporting Information: Study Protocol, SAP, ICF